CLINICAL TRIAL: NCT02564445
Title: Using Social Incentives and Gamification for Weight Loss Promotion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 823326
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Weight Loss; Obesity; Physical Activity
MeSH Terms: conditions — Weight Loss; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Experimental): Participants choose a weight loss goal of 6-8% of baseline weight and given access to a wireless weight scale and smartphone application activity tracker to receive feedback on weight and feedback on step counts.
  They will be given information on the federal and CDC guidelines for physical activity and will also be told that they should strive to achieve 10,000 steps per day to help promote weight loss.
  Interventions: Behavioral: Feedback on weight; Behavioral: Feedback on step counts
- Gamification (Experimental): Participants choose a weight loss goal of 6-8% of baseline weight and given access to a wireless weight scale and smartphone application activity tracker to receive feedback on weight and feedback on step counts.
  All participants play a game with their teammate that includes points, levels and the opportunity to win a trophy, plaque or medal. They will advance or not advance based on their progress with weight loss and physical activity through 24 weeks. During the 12-week follow-up they'll be asked to maintain or make progress toward their weight loss goal.
  Interventions: Behavioral: Gamification; Behavioral: Feedback on weight; Behavioral: Feedback on step counts
- Gamification + Share Data with PCP (Experimental): Participants choose a weight loss goal of 6-8% of baseline weight and given access to a wireless weight scale and smartphone application activity tracker to receive feedback on weight and feedback on step counts.
  Participants will be asked to allow the study team to share their weight and step data with their primary care physician (PCP).
  All participants play a game with their teammate that includes points, levels and the opportunity to win a trophy, plaque or medal. They will advance or not advance based on their progress with weight loss and physical activity through 24 weeks. During the 12-week follow-up they'll be asked to maintain or make progress toward their weight loss goal.
  Interventions: Behavioral: Gamification; Behavioral: Share Data with PCP; Behavioral: Feedback on weight; Behavioral: Feedback on step counts

INTERVENTIONS:
Behavioral: Gamification — All participants will be entered with their teammate into a game that includes points and levels
  Arms: Gamification; Gamification + Share Data with PCP
Behavioral: Share Data with PCP — Weight and step count data will be shared with the participant's primary care physician
  Arms: Gamification + Share Data with PCP
Behavioral: Feedback on weight — Participants will use a wireless weight scale to weigh-in at home and receive feedback on weight.
Behavioral: Feedback on step counts — Participants will use a smartphone application that uses accelerometers within the phone to track step counts and receive feedback on step counts

SUMMARY:
This is a 36-week, three-arm randomized, controlled trial using a team-based model to compare two weight loss programs to control. Each intervention will use insights from behavioral economics to leverage social incentives and gamification.

DETAILED DESCRIPTION:
Obesity is a leading risk factor for morbidity and mortality affecting more than one in three adults in the United States. Modifiable health behaviors contribute to this growing epidemic. Insights from behavioral economics have shown promise for motivating behavior change through the use of financial incentives. However, social incentives or those influences that impact individuals to adjust their inherent behaviors based on social ties and connections have not been well examined. Social incentives are a more patient-centered approach that leverages and enhances the existing connections and influences on the individual. Since one individual's behavior change is connected to many others within their network, social incentives have the potential to be a scalable intervention that impacts the community. Gamification, or the use of game design in non-game situations, is often used in the real world, but its effectiveness is unknown. In this study, investigators will conduct a 36-week, three-arm, randomized, controlled trial using a team-based model to compare two weight loss programs to control. Each intervention will use insights from behavioral economics to leverage social incentives and gamification.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Ability to read and provide informed consent
* Has an iPhone 4 or newer
* Have self-reported body mass index of 30 or greater and in-person body mass index of 28 or greater

Exclusion Criteria:

* Conditions that would make participation infeasible such as inability to provide informed consent, illiteracy or inability to speak, read, and write English
* Conditions that would make participation unsafe such as current treatment for drug or alcohol use, myocardial infarction or stroke within the last 6 months, metastatic cancer, pregnant, breastfeeding or plan to become pregnant during study period, previous diagnosis of an eating disorder, or history of unsafe weight loss practices
* Already enrolled in another weight loss study
* Any other medical conditions or reasons that they could not complete a 36-week weight loss program

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in weight in pounds | 24-week primary intervention period

SECONDARY OUTCOMES:
Change in weight in pounds | 12-week follow-up period
Physical activity (mean daily steps) | 24-week primary intervention period
Physical activity (mean daily steps) | 12-week follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Patel, MD, MBA, MS, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No